CLINICAL TRIAL: NCT01312233
Title: Co-Management of Older Adults With Low Back Pain by Medical Physicians and Doctors of Chiropractic
Brief Title: Collaborative Care for Older Adults With Back Pain (COCOA)
Acronym: COCOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Genesis Family Medical Center (Unknown); University of Iowa (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R18HP15126-02
Record Dates: First submitted 2011-03-04; First posted 2011-03-10 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical Care (Active Comparator): Conventional medical care alone
  Interventions: Other: Medical Care
- Dual Care (Active Comparator): Unlinked co-occurrence of conventional medical care and chiropractic care
  Interventions: Other: Dual Care
- Shared Care (Active Comparator): Co-management of medical care and chiropractic care
  Interventions: Other: Shared Care

INTERVENTIONS:
Other: Medical Care — Participants allocated to all three treatment groups receive medical care over a 12-week period. Medical treatments are standard therapies for back pain. Medical and osteopathic physicians follow clinical practice guideline recommendations for back pain: focused history and physical exam; limited diagnostic imaging; self-management education; maintaining physical activity as tolerated and local heat/cold application; pharmacotherapy with analgesics and anti-inflammatory agents. Participants not responding to treatment may receive additional therapies such as physical therapy or specialist referral.
  Other Names: Standard Medical Therapies for Back Pain
  Arms: Medical Care
Other: Dual Care — Participants allocated to Dual Care receive medical care as described plus chiropractic care over a 12-week period. Chiropractic care includes standard therapies for back pain. A doctor of chiropractic determines the therapeutic approach based upon a participant's clinical presentation. Treatments may include spinal or extremity joint manipulation, such as: high velocity-low amplitude or low velocity-variable amplitude maneuvers; mechanical device assisted adjustments; or passive mobilization. Recommendations for exercise, lifestyle modifications, or other therapies may be provided.
  Other Names: Medical Care Plus Chiropractic Care
  Arms: Dual Care
Other: Shared Care — Participants allocated to Shared Care receive co-managed medical care from a medical or osteopathic doctor and chiropractic care from a doctor of chiropractic over a 12-week period. The medical and chiropractic treatments are standard therapies for back pain, as described under Medical Care and Dual Care.
  Other Names: Co-managed Medical Care and Chiropractic Care
  Arms: Shared Care

SUMMARY:
The purpose of the Collaborative Care for Older Adults with Back Pain (COCOA) Clinical Trial is to evaluate the clinical effectiveness and feasibility of a collaborative care model (medical and chiropractic care) through a pragmatic, prospective pilot trial conducted with 120 older adults over the age of 65 with low back pain of at least 1 month duration.

DETAILED DESCRIPTION:
As America ages, cost-effective care for chronic diseases, such as low back pain, becomes more important. Although estimates vary, 70-85% of Americans will suffer from back pain at some point in their lives. Back pain is well established as one of the most common reasons for seeking care from a medical doctor. The American public also turns to alternative medicine providers, such as doctors of chiropractic, for back pain care. However, few clinical examples and little scientific evidence exist of care coordination between these two provider groups in general, and none that specifically target older adults above the age of 65. The purpose of the Collaborative Care for Older Adults with Back Pain (COCOA) Clinical Trial is to evaluate the clinical effectiveness and feasibility of a collaborative care model (medical and chiropractic care) through a pragmatic, prospective pilot trial conducted with 120 older adults over the age of 65 with low back pain of at least 1 month duration. Participants will be randomized to 3-parallel treatment arms: a) conventional medical care (MED CARE), b) unlinked conventional medical and chiropractic care (DUAL CARE), and c) a co-management model including conventional medical and chiropractic care (SHARED CARE). Participants in all three groups will receive up to 12 weeks of usual back pain treatment from medical doctors or doctors of osteopathy (MD/DO) at Genesis Family Medical Center. Participants in two treatment groups additionally will receive up to 12 weeks of usual chiropractic care for back pain from doctors of chiropractic at the Palmer Research Clinic. Outcomes including pain, disability and secondary outcomes will be measured at 1, 2, and 3 months (primary endpoint) with follow-up assessments completed by telephone at 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Low back pain ≥4 on the 11-point Numerical Rating Scale
* Low back pain diagnosis consistent with Quebec Task Force (QTF) Classifications 1-9
* Ambulatory mobility status per successful completion of the Timed Up & Go Test
* Willingness to participate in this clinical trial regardless of treatment group assignment

Exclusion Criteria:

* No history or current episode of low back pain
* Low back pain duration of less than 1 month
* Low back pain diagnosis consistent with Quebec Task Force Classification of 10 or 11
* Any healthcare provider treatment for low back pain in past 2 months
* Currently seeking or receiving compensation for a work-related injury or personal injury case for low back pain
* Currently seeking or applying for disability payments for any health condition
* Spine or neck surgery in the past 3 months
* Broken bone in any location in the body in the past 6 weeks
* Active carcinoma/metastatic disease or current treatment for any form of cancer
* Aortic aneurysm (or suspicion of) >5cm
* Serious concomitant illness or co-morbidity
* Alcohol or drug abuse or dependence
* Need for laboratory testing, diagnostic imaging beyond plain film x-rays or referral to a healthcare provider not associated with the study to determine a diagnosis or for necessary treatment
* Activities of daily living (ADL), mobility impairment or sensory impairment that impacts safety
* Cognitive or memory impairment
* Compliance concerns
* Nursing home residence
* No reliable transportation
* Plans to move from Quad-Cities in the next 4 months
* Pregnancy or plans to become pregnant in next 4 months in a female participant
* Enrollment in this study by another individual who currently lives in the same household as the participant
* Inability to speak (verbally comprehend), read or write in English language
* Unwillingness to avoid all forms of low back pain treatment from non-study medical doctors and chiropractors during study participation
* Unwillingness to enroll in clinical trial regardless of treatment group assignment
* Unwillingness to sign informed consent document
* Current student, employee or faculty member of the Palmer College of Chiropractic or Genesis Family Medical Center

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Goertz, DC, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (2):
- United States (2):
  - Genesis Family Medical Center, Davenport, Iowa
  - Palmer College of Chiropractic, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No
Feasibility/pilot study

REFERENCES:
- [Background] Goertz CM, Salsbury SA, Vining RD, Long CR, Andresen AA, Jones ME, Lyons KJ, Hondras MA, Killinger LZ, Wolinsky FD, Wallace RB. Collaborative Care for Older Adults with low back pain by family medicine physicians and doctors of chiropractic (COCOA): study protocol for a randomized controlled trial. Trials. 2013 Jan 16;14:18. doi: 10.1186/1745-6215-14-18. PMID 23324133
- [Background] Vining RD, Salsbury SA, Pohlman KA. Eligibility determination for clinical trials: development of a case review process at a chiropractic research center. Trials. 2014 Oct 24;15:406. doi: 10.1186/1745-6215-15-406. PMID 25344427
- [Background] Goertz C, Lyons SS, Andresen A, Hondras M, Jones M, Killinger LZ, Long C, Lyons K, Mulhausen P, Vining R. Collaborative Care for Older Adults (COCOA), Palmer College of Chiropractic. J Allied Health. 2010 Fall;39 Suppl 1:e135-6. PMID 21174032
- [Background] Lyons KJ, Salsbury SA, Hondras MA, Jones ME, Andresen AA, Goertz CM. Perspectives of older adults on co-management of low back pain by doctors of chiropractic and family medicine physicians: a focus group study. BMC Complement Altern Med. 2013 Sep 16;13:225. doi: 10.1186/1472-6882-13-225. PMID 24040970
- [Background] Seidman MB, Vining RD, Salsbury SA. Collaborative care for a patient with complex low back pain and long-term tobacco use: a case report. J Can Chiropr Assoc. 2015 Sep;59(3):216-25. PMID 26500355
- [Background] Boysen JC, Shannon ZK, Khan YA, Wells BM, Vining RD. A graphical clinical decision aid for managing imaging report information. J Chiropr Educ. 2017 Mar;32(1):43-49. doi: 10.7899/JCE-17-6. Epub 2017 Dec 19. PMID 29257708
- [Background] Salsbury SA, Goertz CM, Vining RD, Hondras MA, Andresen AA, Long CR, Lyons KJ, Killinger LZ, Wallace RB. Interdisciplinary Practice Models for Older Adults With Back Pain: A Qualitative Evaluation. Gerontologist. 2018 Mar 19;58(2):376-387. doi: 10.1093/geront/gnw188. PMID 28082277
- [Background] Salsbury SA, Vining RD, Hondras MA, Wallace RB, Lyons KJ, Killinger LZ, Goertz CM. Interprofessional Attitudes and Interdisciplinary Practices for Older Adults With Back Pain Among Doctors of Chiropractic: A Descriptive Survey. J Manipulative Physiol Ther. 2019 May;42(4):295-305. doi: 10.1016/j.jmpt.2018.11.011. Epub 2019 Jun 27. PMID 31257002
- [Background] Wells BM, Salsbury SA, Nightingale LM, Derby DC, Lawrence DJ, Goertz CM. Improper Communication Makes for Squat: A Qualitative Study of the Health-Care Processes Experienced By Older Adults in a Clinical Trial for Back Pain. J Patient Exp. 2020 Aug;7(4):507-515. doi: 10.1177/2374373519860347. Epub 2019 Jul 8. PMID 33062871
- [Result] Goertz CM, Salsbury SA, Long CR, Vining RD, Andresen AA, Hondras MA, Lyons KJ, Killinger LZ, Wolinsky FD, Wallace RB. Patient-centered professional practice models for managing low back pain in older adults: a pilot randomized controlled trial. BMC Geriatr. 2017 Oct 13;17(1):235. doi: 10.1186/s12877-017-0624-z. PMID 29029606
- See also: Collaborative care for a patient with complex low back pain and long-term tobacco use: a case report — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4593044/
- See also: Eligibility determination for clinical trials: development of a case review process at a chiropractic research center — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4221721/
- See also: Collaborative Care for Older Adults with low back pain by family medicine physicians and doctors of chiropractic (COCOA): study protocol for a randomized controlled trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3557195/
- See also: Perspectives of older adults on co-management of low back pain by doctors of chiropractic and family medicine physicians: a focus group study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3847523/
- See also: Patient-centered professional practice models for managing low back pain in older adults: a pilot randomized controlled trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5640949/
- See also: Improper communication makes for squat: a qualitative study of the health-care processes experienced by older adults in a clinical trial for back pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7534140/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shared Care | Dual Care | Medical Care
Started | 44 | 44 | 43
Completed | 42 | 44 | 36
Not Completed | 2 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shared Care | Dual Care | Medical Care | Total
Number analyzed (Participants) | 44 | 44 | 43 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (6.2) | 72.3 (6.0) | 72.7 (6.4) | 72.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 19 | 51
  Male | 28 | 28 | 24 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 40 | 43 | 40 | 123
  Race: Other | 4 | 1 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 43 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-Rated Low Back Pain (LBP), an 11 Point Numerical Rating Scale (NRS)
Description: Adjusted mean changes in patient-rated LBP from baseline to week 12 were assessed. Average and worst LBP were rated on an 11 Numerical Rating Scale (NRS) point scale (0, no LBP; 10 worst LBP possible)
Time Frame: Baseline and 3 months
Population: 9 participants (shared care, n=2 / Med Care n=7) did not complete the 3 month appointment due to either withdrawal or loss to follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shared Care | Dual Care | Medical Care
Number analyzed (Participants) | 42 | 44 | 36
units on a scale
  NRS - Average LBP (adjusted mean change) | 1.8 [1.0 to 2.6] | 3.0 [2.3 to 3.8] | 2.3 [1.5 to 3.2]
  NRS - Worst LBP (adjusted mean change) | 2.1 [1.3 to 2.9] | 2.9 [2.1 to 3.6] | 2.3 [1.5 to 3.1]

2. Primary Outcome: Change From Baseline in Patient-Rated Disability, the 24-item Roland Morris Disability Questionnaire (RMDQ)
Description: Adjusted mean changes in patient-rated disability from baseline to week 12 were assessed using the 24-item RMDQ where 0 indicated no disability and 24 indicated severe disability.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shared Care | Dual Care | Medical Care
Number analyzed (Participants) | 42 | 44 | 36
units on a scale | 2.8 [1.6 to 4.0] | 2.5 [1.3 to 3.7] | 1.5 [0.2 to 2.8]

3. Secondary Outcome: Veterans-RAND 36-item Short-Form Health Survey (VR-36)
Description: Physical function and Emotional Well-being (range 0-100). Higher scores indicate a better outcome.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Shared Care | Dual Care | Medical Care
Number analyzed (Participants) | 42 | 44 | 36
units on a scale (0-100)
  Physical Function - Baseline | 50.0 (26.9) | 57.8 (23.6) | 65.0 (23.3)
  Physical Function - 3 Months | 58.8 (26.2) | 63.8 (25.4) | 65.6 (24.2)
  Emotional Well-Being - Baseline | 78.5 (13.1) | 80.4 (14.0) | 77.8 (13.3)
  Emotional Well-Being - 3 Months | 80.9 (14.1) | 82.4 (12.4) | 82.2 (12.9)

4. Secondary Outcome: Change From Baseline in Bothersomeness of Low Back Pain Symptoms
Description: Adjusted mean changes in patient-reported LBP bothersomeness on a 5 point scale index (1, not at all bothered; 5, extremely bothered) from baseline to week 12 were assessed.
Time Frame: Baseline to 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shared Care | Dual Care | Medical Care
Number analyzed (Participants) | 42 | 44 | 36
units on a scale | 0.8 [0.4 to 1.1] | 0.9 [0.6 to 1.2] | 0.6 [0.3 to 0.9]

5. Secondary Outcome: Patient Satisfaction With Care
Description: Percent of participants reporting levels of satisfaction for the information received regarding the cause of low back pain [LBP] (A), prognosis of LBP (B) and activities that hasten recovery (C), concern of MDs and Doctor of Chiropractic (DCs) during treatments (D), the quality of the treatment recommendations(E) and the overall care for LBP (F)
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Shared Care | Dual Care | Medical Care
Number analyzed (Participants) | 42 | 44 | 36
Participants
  (A) Cause of LBP: Poor | 1 | 0 | 7
  (A) Cause of LBP: Fair | 2 | 2 | 4
  (A) Cause of LBP: Good | 10 | 7 | 8
  (A) Cause of LBP: Very Good | 12 | 14 | 15
  (A) Cause of LBP: Excellent | 17 | 21 | 2
  (B) Prognosis of LBP: Poor | 0 | 0 | 6
  (B) Prognosis of LBP: Fair | 5 | 1 | 7
  (B) Prognosis of LBP: Good | 10 | 10 | 6
  (B) Prognosis of LBP: Very Good | 14 | 15 | 16
  (B) Prognosis of LBP: Excellent | 13 | 18 | 1
  (C) Activities that hasten recovery: Poor | 0 | 0 | 5
  (C) Activities that hasten recovery: Fair | 2 | 1 | 6
  (C) Activities that hasten recovery: Good | 10 | 8 | 8
  (C) Activities that hasten recovery: Very Good | 12 | 11 | 14
  (C) Activities that hasten recovery: Excellent | 18 | 24 | 3
  (D) Concern of MDs and DCs during recovery: Poor | 1 | 0 | 2
  (D) Concern of MDs and DCs during recovery: Fair | 1 | 0 | 2
  (D) Concern of MDs and DCs during recovery: Good | 6 | 1 | 8
  (D) Concern of MDs and DCs during recovery: Very Good | 7 | 7 | 11
  (D) Concern of MDs and DCs during recovery: Excellent | 27 | 36 | 13
  (E) Quality of treatment recommendations: Poor | 0 | 0 | 3
  (E) Quality of treatment recommendations: Fair | 0 | 1 | 5
  (E) Quality of treatment recommendations: Good | 6 | 2 | 8
  (E) Quality of treatment recommendations: Very Good | 11 | 11 | 12
  (E) Quality of treatment recommendations: Excellent | 25 | 30 | 8
  (F) Overall Care for LBP: Poor | 0 | 0 | 4
  (F) Overall Care for LBP: Fair | 1 | 0 | 7
  (F) Overall Care for LBP: Good | 5 | 4 | 4
  (F) Overall Care for LBP: Very Good | 14 | 8 | 17
  (F) Overall Care for LBP: Excellent | 22 | 32 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
Arm/Group | Shared Care | Dual Care | Medical Care
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 34/44 | 36/44 | 10/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shared Care (N=44) | Dual Care (N=44) | Medical Care (N=43)
Spine-related pain (Musculoskeletal and connective tissue disorders) | 29 (80) | 33 (118) | 2 (3)
Spine-related pain with radiation (Musculoskeletal and connective tissue disorders) | 7 (10) | 11 (19) | 3 (3)
Extremity pain (Musculoskeletal and connective tissue disorders) | 11 (16) | 18 (35) | 1 (2)
Headache (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0)
General stiffness/tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle spasm/cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Numbness/tingling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
General soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tiredness/fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness/imbalance/vertigo (General disorders) | 4 (6) | 0 (0) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (General disorders) | 5 (5) | 2 (3) | 1 (1)
Lower respiratory infection (General disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion/respiratory symptoms/allergy (General disorders) | 4 (4) | 4 (4) | 0 (0)
Migraine (General disorders) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Laceration (General disorders) | 2 (2) | 6 (7) | 0 (0)
Swelling (General disorders) | 1 (2) | 2 (2) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 3 (3) | 0 (0)
General soreness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chipped tooth (General disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sore (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 4 (5) | 6 (6) | 1 (1)
Skin burning sensation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (General disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (General disorders) | 1 (1) | 0 (0) | 0 (0)
GERD (General disorders) | 0 (0) | 1 (1) | 0 (0)
Skin allergic reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (General disorders) | 0 (0) | 1 (1) | 0 (0)
Concussion (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes